CLINICAL TRIAL: NCT01623115
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of SAR236553/REGN727 in Patients With Heterozygous Familial Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Brief Title: Efficacy and Safety of Alirocumab (SAR236553/REGN727) Versus Placebo on Top of Lipid-Modifying Therapy in Patients With Heterozygous Familial Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Acronym: ODYSSEY FH I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC12492; U1111-1121-4275 (Other: UTN); 2011-005109-56 (EudraCT Number)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Hypercholesterolemia
Keywords: PCSK9
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo for alirocumab every 2 weeks (Q2W) on top of stable lipid-modifying therapy (LMT) for 78 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Lipid Modifying Therapy (LMT)
- Alirocumab 75 mg/Up to 150 mg Q2W (Experimental): Alirocumab 75 mg Q2W on top of stable LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥ 70 mg/dL (1.81 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Lipid Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Alirocumab — Solution for subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre filled pen).
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab 75 mg/Up to 150 mg Q2W
Drug: Placebo (for alirocumab) — Solution for subcutaneous injection in the abdomen, thigh, or outer area of the upper arm by self-injection or by another designated person using auto-injector (also known as pre filled pen).
  Arms: Placebo
Drug: Lipid Modifying Therapy (LMT) — Statin (rosuvastatin, simvastatin or atorvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Alirocumab (SAR236553/REGN727) is a fully human monoclonal antibody that binds PCSK9 (proprotein convertase subtilisin/kexin type 9).

Primary Objective of the study:

To evaluate the effect of alirocumab on low-density lipoprotein cholesterol (LDL-C) levels after 24 weeks of treatment in comparison with placebo.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with placebo on LDL-C at other time points
* To evaluate the effects of alirocumab on other lipid parameters
* To evaluate the safety and tolerability of alirocumab

DETAILED DESCRIPTION:
The maximum study duration was planned to be 89 weeks per participant including participants who successfully completed the 78-week treatment period had the possibility to join an open-label extension study (LTS13463, NCT01954394) at the end of the treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with heterozygous familial hypercholesterolemia who were not adequately controlled with their lipid-modifying therapy

Exclusion criteria:

* Age < 18 years or legal age of adulthood, whichever is greater
* LDL-C < 70 mg/dL (1.81 mmol/L) and with cardiovascular disease
* LDL-C < 100 mg/dL (2.59 mmol/L) and without cardiovascular disease
* Fasting serum triglycerides > 400 mg/dL (4.52 mmol/L)
* Known history of homozygous familial hypercholesterolemia

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (91):
- United States (26):
  - Investigational Site Number 840417, Bell Gardens, California
  - Investigational Site Number 840429, Long Beach, California
  - Investigational Site Number 840419, Los Angeles, California
  - Investigational Site Number 840421, Mission Viejo, California
  - Investigational Site Number 840412, Newport Beach, California
  - Investigational Site Number 840428, Newport Beach, California
  - Investigational Site Number 840461, Northridge, California
  - Investigational Site Number 840452, Washington D.C., District of Columbia
  - Investigational Site Number 840456, Miami, Florida
  - Investigational Site Number 840418, Ponte Vedra, Florida
  - Investigational Site Number 840455, Evanston, Illinois
  - Investigational Site Number 840415, Kansas City, Kansas
  - Investigational Site Number 840425, Auburn, Maine
  - Investigational Site Number 840411, Boston, Massachusetts
  - Investigational Site Number 840409, St Louis, Missouri
  - Investigational Site Number 840407, Morristown, New Jersey
  - Investigational Site Number 840408, New York, New York
  - Investigational Site Number 840401, Charlotte, North Carolina
  - Investigational Site Number 840410, Durham, North Carolina
  - Investigational Site Number 840430, Cincinnati, Ohio
  - Investigational Site Number 840424, Portland, Oregon
  - Investigational Site Number 840404, Philadelphia, Pennsylvania
  - Investigational Site Number 840426, Philadelphia, Pennsylvania
  - Investigational Site Number 840406, Nashville, Tennessee
  - Investigational Site Number 840460, Dallas, Texas
  - Investigational Site Number 840422, Bountiful, Utah
- Austria (3):
  - Investigational Site Number 040403, Graz
  - Investigational Site Number 040402, Vienna
  - Investigational Site Number 040405, Vienna
- Canada (5):
  - Investigational Site Number 124404, Chicoutimi
  - Investigational Site Number 124401, Montreal
  - Investigational Site Number 124403, Québec
  - Investigational Site Number 124406, Sherbrooke
  - Investigational Site Number 124407, Toronto
- Czechia (4):
  - Investigational Site Number 203401, Prague
  - Investigational Site Number 203403, Prague
  - Investigational Site Number 203405, Uherské Hradiště
  - Investigational Site Number 203402, Zlín
- Denmark (2):
  - Investigational Site Number 208401, Copenhagen
  - Investigational Site Number 208403, Esbjerg
- France (3):
  - Investigational Site Number 250403, Dijon
  - Investigational Site Number 250401, Paris
  - Investigational Site Number 250402, Saint-Herblain
- Israel (4):
  - Investigational Site Number 376402, Holon
  - Investigational Site Number 376405, Jerusalem
  - Investigational Site Number 376404, Safed
  - Investigational Site Number 376401, Tel Litwinsky
- Netherlands (8):
  - Investigational Site Number 528406, Amsterdam
  - Investigational Site Number 528410, Amsterdam
  - Investigational Site Number 528408, Den Helder
  - Investigational Site Number 528402, Groningen
  - Investigational Site Number 528411, Leiden
  - Investigational Site Number 528416, Maastricht
  - Investigational Site Number 528409, Nieuwegein
  - Investigational Site Number 528412, Sliedrecht
- Investigational Site Number 578401, Bodø, Norway
- Russia (10):
  - Investigational Site Number 643402, Arkhangelsk
  - Investigational Site Number 643407, Kazan'
  - Investigational Site Number 643409, Moscow
  - Investigational Site Number 643413, Moscow
  - Investigational Site Number 643401, Moscow
  - Investigational Site Number 643412, Novisibirsk
  - Investigational Site Number 643408, Saint Petersburg
  - Investigational Site Number 643406, Saint Petersburg
  - Investigational Site Number 643404, Saint Petersburg
  - Investigational Site Number 643410, Yaroslavl
- South Africa (9):
  - Investigational Site Number 710401, Bloemfontein
  - Investigational Site Number 710405, Bloemfontein
  - Investigational Site Number 710406, Cap Town
  - Investigational Site Number 710402, Cape Town
  - Investigational Site Number 710407, Parktown
  - Investigational Site Number 710403, Parow
  - Investigational Site Number 710408, Pretoria
  - Investigational Site Number 710404, Rondebosch
  - Investigational Site Number 710409, Somerset West
- Spain (9):
  - Investigational Site Number 724403, A Coruña
  - Investigational Site Number 724408, Barcelona
  - Investigational Site Number 724406, Córdoba
  - Investigational Site Number 724407, L'Hospitalet de Llobregat
  - Investigational Site Number 724409, Madrid
  - Investigational Site Number 724401, Madrid
  - Investigational Site Number 724405, Madrid
  - Investigational Site Number 724404, Reus
  - Investigational Site Number 724402, Zaragoza
- Sweden (2):
  - Investigational Site Number 752404, Gothenburg
  - Investigational Site Number 752401, Stockholm
- United Kingdom (5):
  - Investigational Site Number 826402, London
  - Investigational Site Number 826403, London
  - Investigational Site Number 826408, London
  - Investigational Site Number 826409, London
  - Investigational Site Number 826405, Manchester

REFERENCES:
- [Background] Kastelein JJ, Robinson JG, Farnier M, Krempf M, Langslet G, Lorenzato C, Gipe DA, Baccara-Dinet MT. Efficacy and safety of alirocumab in patients with heterozygous familial hypercholesterolemia not adequately controlled with current lipid-lowering therapy: design and rationale of the ODYSSEY FH studies. Cardiovasc Drugs Ther. 2014 Jun;28(3):281-9. doi: 10.1007/s10557-014-6523-z. PMID 24842558
- [Result] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Kastelein JJ, Hovingh GK, Langslet G, Baccara-Dinet MT, Gipe DA, Chaudhari U, Zhao J, Minini P, Farnier M. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 monoclonal antibody alirocumab vs placebo in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Jan-Feb;11(1):195-203.e4. doi: 10.1016/j.jacl.2016.12.004. Epub 2016 Dec 28. PMID 28391886
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 89 centers in 14 countries. A total of 597 participants were screened between July 2012 and April 2013, 111 of whom were screen failures.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction or ischemic stroke, intensity of statin treatment & geographic region. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in 1:2 (placebo:alirocumab) after confirmation of selection criteria. 486 participants were randomized.
Groups:
- Placebo: Placebo for alirocumab subcutaneous (SC) injection every 2 weeks (Q2W) on top of stable lipid-modifying therapy (LMT) for 78 weeks.
- Alirocumab 75 mg/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W on top of stable LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥ 70 mg/dL (1.81 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Started | 163 (Randomized) | 323 (Randomized)
Treated | 163 | 322
Completed | 130 | 246
Not Completed | 33 | 77
Not completed — Randomized but not treated | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Participants moved | 1 | 5
Not completed — Adverse Event | 10 | 13
Not completed — Poor compliance to protocol | 4 | 10
Not completed — Consent withdrawn by participant | 2 | 6
Not completed — Related to study drug administration | 0 | 2
Not completed — Last visit outside protocol visit window | 14 | 26
Not completed — Site closure | 1 | 7
Not completed — Death | 0 | 4
Not completed — Other than specified above | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo for alirocumab SC injection Q2W on top of stable LMT for 78 weeks.
- Alirocumab 75 mg/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W on top of stable LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) at Week 8.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 163 | 323 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (12.3) | 52.1 (12.9) | 51.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 143 | 212
  Male | 94 | 180 | 274
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula (LDL cholesterol = Total cholesterol - HDL cholesterol - [Triglyceride/5]).
  mg/dL | 144.4 (46.8) | 144.8 (51.1) | 144.6 (49.7)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.739 (1.213) | 3.749 (1.325) | 3.746 (1.287)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 9.1 (2.2) | -48.8 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -57.9, 95% CI 2-sided [-63.3 to -52.6] — Alirocumab vs Placebo

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percent change | 8.8 (2.2) | -49.3 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -58.1, 95% CI 2-sided [-63.5 to -52.7] — Alirocumab vs Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 5.7 (2) | -43.5 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -49.2, 95% CI 2-sided [-53.9 to -44.5] — Alirocumab vs Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percent change | 5.7 (2) | -43.9 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -49.5, 95% CI 2-sided [-54.2 to -44.8] — Alirocumab vs Placebo

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 160 | 309
percent change | 4.7 (1.6) | -41.1 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -45.8, 95% CI 2-sided [-49.8 to -41.8] — Alirocumab vs Placebo

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 159 | 308
percent change | 4.5 (1.7) | -41.4 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -45.9, 95% CI 2-sided [-49.9 to -41.8] — Alirocumab vs Placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 9.6 (2) | -42.8 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -52.4, 95% CI 2-sided [-57.2 to -47.6] — Alirocumab vs Placebo

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 52
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percent change | 9.4 (2) | -43.3 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -52.6, 95% CI 2-sided [-57.5 to -47.8] — Alirocumab vs Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 7
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on-or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 7.3 (1.5) | -31.4 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -38.7, 95% CI 2-sided [-42.4 to -35] — Alirocumab vs Placebo

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 160 | 309
percent change | 3.1 (1.5) | -34.5 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -37.5, 95% CI 2-sided [-41.2 to -33.9] — Alirocumab vs Placebo

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 5.3 (1.8) | -38.4 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -43.7, 95% CI 2-sided [-48 to -39.4] — Alirocumab vs Placebo

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 4.1 (1.4) | -28.3 (1)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -32.5, 95% CI 2-sided [-35.7 to -29.2] — Alirocumab vs Placebo

13. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 9 (2.6) | -47.1 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = -56.2, 95% CI 2-sided [-62.4 to -50] — Alirocumab vs Placebo

14. Secondary Outcome: Percentage of Very High Cardiovascular (CV) Risk Participants Achieving Calculated LDL-C < 70 mg/dL (<1.81 mmol/L) or High CV Risk Participants Achieving Calculated LDL-C < 100 mg/dL (<2.59 mmol/L) at Week 24 - ITT Analysis
Description: Very high CV risk participants: Heterozygous Familial Hypercholesterolemia (heFH) participants with coronary heart disease (CHD) or CHD risk equivalents. High CV risk participants: heFH participants without CHD or CHD risk equivalents. CHD risk equivalent: peripheral arterial disease, ischemic stroke, moderate chronic kidney disease (estimated glomerular filtration rate, 30 to <60 ml/minute/1.73 m^2 of body-surface area), or diabetes mellitus plus 2 or more additional risk factors (hypertension; ankle-brachial index of ≤0.90; microalbuminuria, macroalbuminuria, or a urinary dipstick result of >2+ protein; preproliferative or proliferative retinopathy or laser treatment for retinopathy; or a family history of premature CHD). Adjusted percentages at Week 24 were obtained from multiple imputation approach for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percentage of participants | 2.4 | 72.2
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 156, 95% CI 2-sided [48.9 to 498.1] — Alirocumab vs Placebo

15. Secondary Outcome: Percentage of Very High CV Risk Participants Achieving Calculated LDL-C < 70 mg/dL (<1.81 mmol/L) or High CV Risk Participants Achieving Calculated LDL-C < 100 mg/dL (<2.59 mmol/L) at Week 24 - On- Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percentage of participants | 2.4 | 73
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 156.6, 95% CI 2-sided [49.7 to 493.7] — Alirocumab vs Placebo

16. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percentage of participants | 0.8 | 59.8
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 244.9, 95% CI 2-sided [34.4 to 1744.4] — Alirocumab vs Placebo

17. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection.
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percentage of participants | 0.8 | 60.1
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 240, 95% CI 2-sided [33.9 to 1700.7] — Alirocumab vs Placebo

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | -7.5 (2) | -25.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -17.7, 95% CI 2-sided [-22.6 to -12.9] — Alirocumab vs Placebo

19. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 0.8 (1.2) | 8.8 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = 8, 95% CI 2-sided [5 to 11] — Alirocumab vs Placebo

20. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 18
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 6.3 (2.2) | -9.6 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance was ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -16, 95% CI 2-sided [-21.3 to -10.6] — Alirocumab vs Placebo

21. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-1 (Apo A-1) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment (Apo A-1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 160 | 309
percent change | 0.3 (1) | 5 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = 4.7, 95% CI 2-sided [2.3 to 7.2] — Alirocumab vs Placebo

22. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | -3.9 (1.8) | -21.2 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -17.3, 95% CI 2-sided [-21.5 to -13] — Alirocumab vs Placebo

23. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 2.1 (1.2) | 6.4 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = 4.3, 95% CI 2-sided [1.5 to 7.2] — Alirocumab vs Placebo

24. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 22
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 1.7 (2.2) | -8 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0003, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -9.7, 95% CI 2-sided [-15 to -4.4] — Alirocumab vs Placebo

25. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 11
Time Frame: From Baseline to Week 52
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 160 | 309
percent change | 0.1 (1) | 2.9 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0187, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS mean difference = 2.8, 95% CI 2-sided [0.5 to 5.2] — Alirocumab vs Placebo

26. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percent change | 9.1 (2.6) | -48.1 (1.9)

27. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM including all available post-baseline data from Week 4 to Week 78 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 78
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 322
percent change | 11.5 (2.8) | -40.3 (2.0)

28. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 78 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 78 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 78 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 78
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 163 | 321
percent change | 14.0 (2.8) | -43.7 (2.0)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit in the study regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent that is AEs that developed/worsened during the 'treatment-emergent period' (from the first double-blind injection up to the day of the last injection + 70 days or up to first intake in the extension study, whichever came first).
Groups:
- Placebo: Participants exposed to placebo Q2W on top of stable LMT (mean exposure of 72 weeks).
- Alirocumab 75/Up to 150 mg Q2W: Participants exposed to Alirocumab 75 mg/Up to 150 mg Q2W on top of stable LMT (mean exposure of 72 weeks).
Arm/Group | Placebo | Alirocumab 75/Up to 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 22/163 | 44/322
Other Adverse Events (participants affected / at risk) | 70/163 | 142/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Alirocumab 75/Up to 150 mg Q2W (N=322)
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 4
Acute myocardial infarction (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Trousseau's syndrome (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 1
Miscarriage of partner (Social circumstances) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Alirocumab 75/Up to 150 mg Q2W (N=322)
Nasopharyngitis (Infections and infestations) | 12 | 36
Upper respiratory tract infection (Infections and infestations) | 14 | 22
Influenza (Infections and infestations) | 9 | 20
Sinusitis (Infections and infestations) | 7 | 17
Bronchitis (Infections and infestations) | 9 | 10
Headache (Nervous system disorders) | 9 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Injection site reaction (General disorders) | 18 | 40

LIMITATIONS AND CAVEATS:
Manual reclassification was done by the Sponsor for the "other reasons" of non-completion of study as specified in the electronic case report form (eCRF).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.